CLINICAL TRIAL: NCT03097302
Title: Tomographic Analysis of Anterior, Posterior and Total Corneal Refractive Power Changes After Femtosecond Laser-assisted Keratotomy After Laser Lens Surgery
Brief Title: Tomographic Analysis of Anterior, Posterior, Total Corneal Refractive Power Changes After Laser-assisted Keratotomy
Status: Completed | Type: Observational
Sponsor: University Clinic Frankfurt (Other)
Responsible Party: Principal Investigator, Myriam Böhm, Professor Dr. med. Thomas Kohnen, University Clinic Frankfurt
Other Study IDs: 140/13
Record Dates: First submitted 2017-03-18; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Corneal Astigmatism
Keywords: laser-assisted keratotomy; anterior astigmatism; posterior astigmatism; total corneal refractive power; nomogram
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laser keratotomy — Penetrating femtosecond laser assisted keratotomy to treat preexisting corneal astigmatism during lens surgery.

SUMMARY:
To analyze the effect of femtolaser-assisted keratotomy on corneal astigmatism (anterior, posterior and Total corneal refractive power) measured by Scheimpflug tomography after laser lens surgery.

DETAILED DESCRIPTION:
This study investigated patients' eyes with low to moderate total corneal refractive power determined with Scheimpflug tomography (Pentacam HR) after penetrating femtosecond laser-assisted keratotomy (pFLAK) and laser lens surgery. The anterior corneal astigmatism, posterior corneal astigmatism and total corneal refractive power were determined before, 1 month and 3 months after lens surgery. Vector analysis according to the Alpins' method was used to calculate surgically induced astigmatism (SIA).

ELIGIBILITY:
Inclusion Criteria:

- Patients who received penetrating femtosecond laser-assisted lens surgery with low to moderate corneal astigmatism

Exclusion Criteria:

* Eyes with irregular corneal astigmatism such as keratoconus, previous corneal surgery, acute or chronic ophthalmic diseases of the anterior segment and intraoperative complications were not included in this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who received penetrating femtosecond laser-assisted lens surgery with low to moderate corneal astigmatism during lens surgery
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2013-06-06 (Actual); Primary Completion 2014-07-31 (Actual); Study Completion 2014-07-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Total corneal refractive power at 3 months | Before and 3 months after lens surgery
  Total corneal astigmatism (anterior and posterior astigmatism)

SECONDARY OUTCOMES:
Change from Baseline Anterior corneal astigmatism at 3 months | Before and 3 months after lens surgery
  Anterior corneal astigmatism
Change from Baseline Posterior corneal astigmatism at 3 months | Before and 3 months after lens surgery
  Posterior corneal astigmatism

IPD SHARING:
Plan to Share IPD: Yes
Via a Publication in a reviewed journal.